CLINICAL TRIAL: NCT07245173
Title: Randomized Control Trial Comparing the Incidence of Loop Formation in Water Infusion Versus Air Insufflation Colonoscopy Techniques
Brief Title: Randomized Control Trial Comparing the Incidence of Loop Formation in Colonoscopy Techniques
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial University of Newfoundland (Other)
Responsible Party: Principal Investigator, David Pace, Dr. Davis Pace, Memorial University of Newfoundland
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: 41436
Record Dates: First submitted 2025-06-09; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Colon Cancer Screening
MeSH Terms: interventions — Colonoscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colonoscopy with water insufflation (Experimental): Colonoscopy performed using just water to inflate the colon
  Interventions: Diagnostic Test: colonoscopy
- Colonoscopy with air insufflation (Experimental): Colonoscopy performed using just air to inflate the colon
  Interventions: Diagnostic Test: colonoscopy

INTERVENTIONS:
Diagnostic Test: colonoscopy — Colonoscopy performed using just water or just air to inflate the colon

SUMMARY:
A colonoscopy is a common procedure used to check for problems in the colon, such as disease or other health issues. Although it's widely used, one challenge is that the flexible tube used in the procedure (called a colonoscope) can sometimes form loops inside the colon. When this happens, pushing the tube further doesn't help it move forward-it just makes the loop bigger, which can make the procedure harder to complete. These loops can also cause more pain for the patient, require more sedation (medication to relax or put the patient to sleep), and increase the time it takes to finish the procedure. Because of this, it's important to find ways to reduce loop formation. Two common methods used in colonoscopies are called air insufflation and water infusion.

This study will compare the two methods-air vs. water-to see which one causes fewer loops. It will be a randomized controlled trial, meaning participants will be randomly assigned to one of the two methods. The study will involve real patients, and the data will be collected by physicians, residents (doctors in training), and medical students. During the colonoscopies, images from a tool that guides the scope will be recorded on video.

Experienced staff doctors and surgical residents (with at least two months of special training in this procedure) will perform the colonoscopies. Each procedure will be supervised by a team member, such as a medical student, resident, or staff doctor. Afterward, two reviewers who don't know which method was used will watch the videos to look for any loops. They will look for specific types of loops, including n, alpha, reverse alpha, reverse splenic, and gamma loops.

The study will also track how long it takes to reach the end of the colon (called the cecum), how comfortable the patient was (using a standard rating system already used in all colonoscopies), and how much sedation was needed.

ELIGIBILITY:
Inclusion Criteria:

* Consenting patients who are undergoing a routine colonoscopy.
* Ages between 18-80 years old.

Exclusion Criteria:

* Refusal to participate
* Inability to provide informed consent.
* History of prior colonic surgery.
* Poor bowel preparation.
* Known bowel obstruction.
* Emergency colonoscopy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Number and type of colonscopy loops formed | 12 months
  The number and type of different colonoscopy loops formed during each colonoscopy will be recorded from the initial insertion of the colonoscope to complete removal of the colonoscope of each colonoscopy.

IPD SHARING:
Plan to Share IPD: No